CLINICAL TRIAL: NCT00461188
Title: Genetics of Endocrine Tumours - Familial Isolated Pituitary Adenoma - FIPA
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 004842
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Acromegaly; Gigantism; Familial Isolated Pituitary Adenoma; FIPA; Pituitary Adenoma Predisposition; PAP
Keywords: acromegaly; gigantism; familial pituitary adenoma; Familial acromegaly; Familial Isolated Pituitary Adenoma; FIPA; Pituitary adenoma predisposition; PAP
MeSH Terms: conditions — Acromegaly; Gigantism; Pituitary Adenoma, Familial Isolated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA sample, tissue sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The research is aimed at identifying new predisposition genes for endocrine tumours. Our focus initially is on pituitary adenomas including growth hormone-secreting tumors (somatotrophinomas) and prolactin secreting tumours (prolactinomas), but we wish to extend work to other pituitary tumour cases/families.

The recruitment process will be as follows.

1. We will recruit patients from our own Endocrine outpatient clinics and inpatient wards. In addition we will ask colleagues in other Endocrinology Departments (or other specialties such as Clinical Genetics,Pathology, General Medicine ) to identify potentially suitable patients with endocrine & pituitary tumours from their records. We shall focus on patients with good evidence of inheritance of their condition: relatively early onset; or multiple lesions; or other affected family members. Conditions where the predisposing genes have been identified (principally MEN) will be excluded from study. Patients directly contacting us can also enter the study.
2. The Consultant looking after the patient will contact the patient to initially inform him/her of the study.
3. We will then contact the patient (generally by telephone) to discuss the study and what it would entail in terms of information and samples.
4. Subject to agreement in (3), patient will receive 'Information Sheet for patients with pituitary tumour' and 'Consent Form' and will have blood sampling in Consultant's clinic.
5. We will contact additional family members (if appropriate) after an initial approach by the family member already recruited to the study. The additional family members may have developed tumours similar to those of the proband, or may be unaffected individuals who provide useful information for gene identification purposes (for example, spouses may greatly aid the power of gene mapping by linkage. They will receive the "Information Sheet for family members". analysis).

8. Archival tissue will be obtained from HTA licensed tissue banks. This is an established bank whose licence is primarily for diagnosis but can be used for research. 9. We will undertake laboratory work, such as genetic linkage analysis, candidate gene mutation screening and studies of loss of heterozygosity in tumours, to identify the genes predisposing to the condition, such as the AIP gene. In addition we would like to screen other genes related to the chaperon AIP molecule, such as AhR, and other genes currently identified (PDE4A5, survivin and Tom20 protein) or may not been identified.

Blood samples for DNA and RNA will coded with unique ID numbers. Pituitary and other endocrine tumour samples will be collected at surgery and kept in liquid nitrogen or -80 C. They will be coded with unique ID numbers. Candidate gene sequencing will be performed in the Barts and the London Medical School Genome Centre.

RNA expression studies from blood or adenoma tissue samples will be performed by RT-PCR. Protein expression studies will be performed by Western blotting or immunohistochemistry. The first gene we wish to study causes familial acromegaly, a disease resulting from a pituitary adenoma secreting growth hormone.

To establish if the candidate gene is also causing possibly sporadic (not familial) cases of the disease, samples (blood and tissue) will be collected from patients with sporadic disease and will be analysed as above.

DETAILED DESCRIPTION:
We wish to find genes which predispose to pituitary tumours, to find out how those genes work and to assess those genes (and similar genes) in other conditions related to the pituitary tumours.

We will study the recently identified new familial pituitary adenoma gene AIP (AhR interacting protein) and its partner molecules for example AhR (aryl hydrocarbon receptor) in familial and sporadic pituitary adenoma cases.

We have 3 main questions:

Is the identified gene (e.g. AIP) involved in the pathogenesis of familial pituitary tumours (acromegaly), are there any mutations in this gene in these families? What is the function of the new gene in pituitary tumorigenesis? Does the new gene or its partners have a role in sporadic pituitary adenoma tumorigenesis?

Pituitary tumours comprise around 15% of all intracranial neoplasms, and present with distinct clinical characteristics, usually in terms of local space-occupying effects, or secondary to tumoral hypersecretion or its consequences. Acromegaly and gigantism are due in more than 99% of cases to a somatotroph adenoma, which has been demonstrated to be monoclonal in the great majority of instances1. It has been suggested that there are 6 major features of oncogenesis which all need to be present in cases of cancer2, but only 3 of these (activation of an oncogene, inactivation of a tumour suppressor gene [TSG], inhibition of apoptosis) appear to be relevant to pituitary tumorigenesis; these tumours are usually benign adenomas, and the formation of new blood vessels and the capacity for metastasis are uncommon, although some way of evading senescence may be important. It has therefore been suggested that a very small number of mutations in oncogenes and/or TSG's may be causally responsible for pituitary adenomas. This makes them an excellent model for the early stages of tumorigenesis. However, while much has been established regarding the molecular pathology of these tumours, including extensive studies from our own laboratory3-7, the initiating mutation or mutations responsible for tumorigenesis have to date defied analysis.

Early work established that some 30% of patients with acromegaly had one of 2 mutations of the alpha-subunit of the receptor-associated G protein, leading to constitutive activation, but it has been difficult to show that this has relevant biological consequences. We have identified a partial failure of the feedback regulation on somatotroph tumours, but no mutations of the relevant genes have been recorded6,8. We and others have also explored the possibility that there are somatic mutations in sporadic somatotroph tumours of genes identified in some hereditary syndromes associated with acromegaly (MEN-I, Carney syndrome), but these appear to be extremely rare9. However, we have worked in collaboration with a Chicago group who have been seeking to identify the gene responsible for familial acromegaly, a very rare dominant condition10-14. Some 46 families have been described worldwide over the last 40 years, and from a cohort of 8 families a region on chromosome 11q13 has been identified: we have sought to use data from our microarray studies15 to pinpoint the abnormal gene in these patients, but so far unsuccessfully. Our recent work has suggested that there are abnormalities of the cell cycle in pituitary adenomas, especially down-regulation of the cycling-dependent kinase inhibitor p27 and activation of cycling E, and that this is secondary to a putative abnormal growth factor receptor(s), but specific mutations of these receptors are absent16.

Very recently, a Finnish group have identified a dominant gene of very low penetrance which appears to segregate with familial somatotroph and prolactin-secreting tumours17. This lies at or near position 11q13, but it remains unclear as to whether this is indeed the same gene identified in our families with a much more strongly penetrant condition. The gene codes for AIP (= aryl hydrocarbon receptor interacting protein, also known as XAP2 hepatitis B virus X-associated protein 2 or ARA9 = AhR (aryl hydrocarbon receptor)-activated protein 9. AIP has 330 amino acids and has a PPIase-like domain FKBP12 and four tetratricopeptide repeats (TPRs), probably important for protein-protein interactions.

AIP is a putative activating partner for the aryl hydrocarbon receptor, probably increasing the function of AhR. AhR has been linked to the induction of hepatic detoxifying gene products in response to environmental toxins such as dioxin18. However, an additional function appears to be regulation of the cell cycle, suppressing cyclin E and increasing expression of p2719. The AhR also has been shown to interact with cyclic AMP. In this latter instance, the interaction with cAMP appears to compete with the dioxin-dependent pathway, such that AhR has enhanced transport into the nucleus with transcriptional effects quite separate to those stimulated by dioxin and related ligands. As cAMP is an important second messenger in somatotroph tumours, this may be the relevant pathway underlying the apparent activity of AIP as a tumour suppressor.

There is therefore a primary reason to believe that AIP may indeed function as a TSG in pituitary adenomas, and loss of heterozygosity for 11q13 as been seen in tumours in familial cases17. However, the initial Finnish data were only based on 3 families, and we now plan to investigate our entire cohort of families with acromegaly and prolactinomas, as well as further families that we are in the process of collecting. We have contacted many endocrinologists throughout the UK, and we have identified a small number of additional families. Finally, in the initial study some of the patients were apparently isolated cases of acromegaly, but presenting at an unusually young age, especially with gigantism. In such cases too mutations of the AIP gene were recorded.

Plan of Investigation: We plan to screen all known families with a history of acromegaly and/or prolactinomas, as well as other pituitary tumour families to be identified in the UK, for mutations of the AIP gene. In addition we would like to screen other genes related to the chaperon AIP molecule, such as AhR, and other genes currently identified (PDE4A5, survivin and Tom20 protein) or may not been identified. As the data suggest that early onset, aggressive, seemingly sporadic cases of acromegaly or prolactinoma could also be caused by germline mutations, we will include patients with clinically sporadic but early-onset aggressive disease.

The patients will be recruited from Endocrinology Departments from the collaborating centres (Barts Hospital London, Newcastle, Oxford, Stroke-on-Trent, Sheffield, Manchester, Aberdeen and Stroke-on-Trent).

Blood samples will be assessed for germline DNA, RNA and protein isolated for peripheral lymphocytes collected in a peripheral blood sample. Affected family members will be identified, as well as first-degree relatives both affected and unaffected. At the same time, all apparent mutations or polymorphisms of AIP will be tracked in a cohort of 100 germline blood samples from normal volunteers for assessment of the background gene frequency in order to assess their relationship to disease status. Patient tumour samples will collected and RNA and protein expression studied.

ELIGIBILITY:
Inclusion Criteria:

* Familial acromegaly or other type of pituitary tumour OR
* Early onset acromegaly or
* Sporadic pituitary tumour

Exclusion Criteria:

* Do not consent

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pituitary disease patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2007-03-01 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
germline mutation assessment | 10 years
  in selected patient targeted sequencing
SNP genotyping assessment | 10 years
  for all affected subjects

CONTACTS AND LOCATIONS:
Overall Officials: Marta Korbonits, MD PhD, Principal Investigator — Barts and the London Medical School
Locations (3):
- United Kingdom (3):
  - Leicester Infirmary, Leicester
  - Barts and the London medical School, London
  - Royal Victoria Infirmary, Newcastle upon Tyne

REFERENCES:
- [Background] Hernandez-Ramirez LC, Gabrovska P, Denes J, Stals K, Trivellin G, Tilley D, Ferrau F, Evanson J, Ellard S, Grossman AB, Roncaroli F, Gadelha MR, Korbonits M; International FIPA Consortium. Landscape of Familial Isolated and Young-Onset Pituitary Adenomas: Prospective Diagnosis in AIP Mutation Carriers. J Clin Endocrinol Metab. 2015 Sep;100(9):E1242-54. doi: 10.1210/jc.2015-1869. PMID 26186299
- [Background] Iacovazzo D, Caswell R, Bunce B, Jose S, Yuan B, Hernandez-Ramirez LC, Kapur S, Caimari F, Evanson J, Ferrau F, Dang MN, Gabrovska P, Larkin SJ, Ansorge O, Rodd C, Vance ML, Ramirez-Renteria C, Mercado M, Goldstone AP, Buchfelder M, Burren CP, Gurlek A, Dutta P, Choong CS, Cheetham T, Trivellin G, Stratakis CA, Lopes MB, Grossman AB, Trouillas J, Lupski JR, Ellard S, Sampson JR, Roncaroli F, Korbonits M. Germline or somatic GPR101 duplication leads to X-linked acrogigantism: a clinico-pathological and genetic study. Acta Neuropathol Commun. 2016 Jun 1;4(1):56. doi: 10.1186/s40478-016-0328-1. PMID 27245663
- [Background] Radian S, Diekmann Y, Gabrovska P, Holland B, Bradley L, Wallace H, Stals K, Bussell AM, McGurren K, Cuesta M, Ryan AW, Herincs M, Hernandez-Ramirez LC, Holland A, Samuels J, Aflorei ED, Barry S, Denes J, Pernicova I, Stiles CE, Trivellin G, McCloskey R, Ajzensztejn M, Abid N, Akker SA, Mercado M, Cohen M, Thakker RV, Baldeweg S, Barkan A, Musat M, Levy M, Orme SM, Unterlander M, Burger J, Kumar AV, Ellard S, McPartlin J, McManus R, Linden GJ, Atkinson B, Balding DJ, Agha A, Thompson CJ, Hunter SJ, Thomas MG, Morrison PJ, Korbonits M. Increased Population Risk of AIP-Related Acromegaly and Gigantism in Ireland. Hum Mutat. 2017 Jan;38(1):78-85. doi: 10.1002/humu.23121. Epub 2016 Oct 4. PMID 27650164
- [Background] Caimari F, Hernandez-Ramirez LC, Dang MN, Gabrovska P, Iacovazzo D, Stals K, Ellard S, Korbonits M; International FIPA consortium. Risk category system to identify pituitary adenoma patients with AIP mutations. J Med Genet. 2018 Apr;55(4):254-260. doi: 10.1136/jmedgenet-2017-104957. Epub 2018 Feb 10. PMID 29440248
- [Background] Marques P, Caimari F, Hernandez-Ramirez LC, Collier D, Iacovazzo D, Ronaldson A, Magid K, Lim CT, Stals K, Ellard S, Grossman AB, Korbonits M; FIPA Consortium. Significant Benefits of AIP Testing and Clinical Screening in Familial Isolated and Young-onset Pituitary Tumors. J Clin Endocrinol Metab. 2020 Jun 1;105(6):e2247-60. doi: 10.1210/clinem/dgaa040. PMID 31996917
- [Result] Chahal HS, Stals K, Unterlander M, Balding DJ, Thomas MG, Kumar AV, Besser GM, Atkinson AB, Morrison PJ, Howlett TA, Levy MJ, Orme SM, Akker SA, Abel RL, Grossman AB, Burger J, Ellard S, Korbonits M. AIP mutation in pituitary adenomas in the 18th century and today. N Engl J Med. 2011 Jan 6;364(1):43-50. doi: 10.1056/NEJMoa1008020. PMID 21208107
- [Derived] Hernandez-Ramirez LC, Martucci F, Morgan RM, Trivellin G, Tilley D, Ramos-Guajardo N, Iacovazzo D, D'Acquisto F, Prodromou C, Korbonits M. Rapid Proteasomal Degradation of Mutant Proteins Is the Primary Mechanism Leading to Tumorigenesis in Patients With Missense AIP Mutations. J Clin Endocrinol Metab. 2016 Aug;101(8):3144-54. doi: 10.1210/jc.2016-1307. Epub 2016 Jun 2. PMID 27253664
- See also: This website describes the main characteristics of Familial Isolated Pituitary Adenoma (FIPA) — http://www.fipapatients.org/

DOCUMENTS (1):
  • Study Protocol (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT00461188/Prot_000.pdf